CLINICAL TRIAL: NCT07016022
Title: Variability and Post-op AEs: Does Preoperative CardioPulmonary Variability Assessment Identify Risk of Postoperative Adverse Events Following Thoracic Surgery
Acronym: CPVA
Status: Not yet recruiting | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20250214-01H
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Thoracic Cancer; Complication,Postoperative
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CardioPulmonary Variability Assessment — The Preoperative CardioPulmonary Variability Assessment (CPVA) will assess baseline HRV & RRV and the ability to tolerate mild physiologic stress. The assessment will involve a a Philips MP50 monitor that will collect continuous ECG (Lead II) and CO2-based respiratory waveform data with intermittent blood pressure (BP) measurements over a test of less than 60 minutes. We will measure the response to mild physiological stress which reflects adaptability, autonomic function and functional mobility by having the participant perform certain tasks such as sitting, standing, deep breathing, valsalva manoeuvres, and marching.

SUMMARY:
Major thoracic surgery is high risk as it carries a significant risk of postoperative Adverse Events (AEs), where patients experience complications and do not recover as expected. These AEs can increase the risk of mortality, hospital length of stay, as well as healthcare costs. The investigators' aim is to improve surgical safety by pioneering a marked advance in preoperative prediction of postoperative AEs that will enable individualized targeted perioperative pathways to prevent postoperative AEs. Given that illness and stress are associated with a loss in physiologic variability (e.g. heart and respiration rate), the investigators will use heart and lung variability assessments to improve prediction of postoperative AEs. Therefore, this study aims to assess the feasibility of implementing a preoperative CardioPulmonary variability assessment; determine if preoperative CardioPulmonary variability is associated with postoperative AEs; and determine if this variability assessment is superior and complementary to existing measures of risk and frailty.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years of age)
* Patients undergoing major thoracic resection for lung, esophageal or gastric cancer or mediastinal tumour (at least lobectomy, pneumonectomy, esophagectomy, gastrectomy, or mediastinal tumour resection)

Exclusion Criteria:

* Urgent/emergent cases
* Patients with pre-existing atrial fibrillation or arrhythmia (persistent/paroxysmal)
* Patients that are pacemaker dependent
* Patients unable to participate in preoperative testing protocol (CardioPulmonary Variability Assessment)
* Patients that are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing major thoracic surgery who have no history of atrial fibrillation or arrhythmia, are not pacemaker dependent, and are not pregnant.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of implementing CPVA testing in thoracic surgery patients | Upon study completion, 10 months after study initiation
  Implementing CPVA testing in thoracic surgery patients will be considered feasible if:
  >50% of identified eligible patients are enrolled and consented, >90% of consented and enrolled patients complete CPVA testing protocol There is adequate data analysis from the CPVA in >90% of patients that complete the CPVA protocol >95% of CRFs are complete
Statistical association between preoperative HRV and RRV and major cardiac and pulmonary postoperative AEs | Upon study completion, 10 months after study initiation
  The statistical association between preoperative HRV and RRV and major cardiac and pulmonary postoperative AEs will be determined by separating the patient's into subgroups based on (a) any AEs (any class), (b) serious AEs (Class III and above), (c) the type of AEs they experience (including POPCs, atrial fibrillation, air leak) and performing statistical analyses to determine if there is a significance between patients who experience AEs and those who don't based on the CPVA metrics.

SECONDARY OUTCOMES:
Assess predictive power of CPVA indices | Upon study completion, 10 months after study initiation
  A simple univariate logistic regression model will be created for each variability metric and literature-based thresholds will be used for the CPVA indices to assess their predictive power, which will be compared to that of the current predictor for the 3 types of AEs (POPC, arrhythmia, air leak). For each AE, a multiple logistic regression using the original predictors and variability features will also be performed to assess the added value of the variability features.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew JE Seely, MD, PhD, FRSCS, Principal Investigator — The Ottawa Hospital

IPD SHARING:
Plan to Share IPD: No